CLINICAL TRIAL: NCT06342388
Title: Enrollment Barriers, Procedural Denials, and Loss of Medicaid Coverage: A Randomized Trial to Identify and Implement Effective Outreach Solutions
Brief Title: Enrollment Barriers, Procedural Denials, and Loss of Medicaid Coverage
Status: Withdrawn | Type: Observational
Why Stopped: Record created in error.
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Covering Wisconsin (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2024-0427; A538500 (Other: UW- Madison); Protocol Version 3/20/2024 (Other: UW- Madison); SMPH/POP HEALTH SCI/POP HLTH (Other: UW- Madison)
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: No Medicaid Coverage
Keywords: Medicaid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Live Outreach: People in this cohort will receive a live outbound call from a Navigator
- Pre-recorded Outreach: People in this cohort will receive a pre-recorded outbound call providing a hotline number
- No outreach: People in this cohort will not receive outreach of any kind

SUMMARY:
The goal of this study is to try new outreach methods to improve access to Medicaid for those who lost Medicaid for procedural reasons. The main questions it aims to answer are:

1. How does a live phone call from a Navigator impact Medicaid enrollment among people who lost Medicaid coverage for procedural reasons?
2. What is the effectiveness of outreach using a live call rather than a pre-recorded call?

ELIGIBILITY:
Inclusion Criteria:

* Eligible for Medicaid
* Lost Medicaid coverage between June 2024 and November 2025

Exclusion Criteria:

* Preferring a language other than English, Spanish, or Hmong
* No working phone number

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: People in Wisconsin who lost Medicaid coverage for procedural reasons any time between June 2024 and November 2025
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-07 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of people who successfully renew their Medicaid coverage within 3 months of receiving the live outbound call | 3 months
  Numbers will be counted using Wisconsin administrative data on Medicaid enrollment housed at the UW Institute for Research on Poverty.

SECONDARY OUTCOMES:
Duration of coverage gaps | 6 months
  Duration of gaps will be measured using Wisconsin administrative data on Medicaid enrollment housed at the UW Institute for Research on Poverty.
Number of people who successfully renew their Medicaid coverage within 6 months of receiving the live outbound call | 6 months
  Numbers will be counted using Wisconsin administrative data on Medicaid enrollment housed at the UW Institute for Research on Poverty.
Number of people who successfully renew their Medicaid coverage within 6 months of receiving the pre-recorded outbound call | 6 months
  Numbers will be counted using Wisconsin administrative data on Medicaid enrollment housed at the UW Institute for Research on Poverty.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Myerson, PhD, Principal Investigator — University of Wisconsin, Madison

IPD SHARING:
Plan to Share IPD: No